CLINICAL TRIAL: NCT05527860
Title: Evolution of the State of Health of Patients Undergoing Surgery for Osteoarticular Surgery: Retrospective Study Based on the Point of View of Patients
Brief Title: Evolution of the State of Health of Patients Undergoing Surgery for Osteoarticular Surgery
Acronym: EPOPEE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8580
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Chronic pain; Osteoarticular surgery
MeSH Terms: conditions — Osteoarthritis; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteoarticular surgery is frequently associated with the occurrence of moderate to severe postoperative pain. This pain can persist and become chronic post-surgical pain that is often debilitating. The transition between early postoperative pain and chronic pain is poorly understood, which complicates treatment.

ELIGIBILITY:
Inclusion criteria:

* Patient aged ≥18 years
* Underwent osteoarticular surgery between 01/01/2019 and 31/12/2022.
* Having been followed up with the administration of at least 1 QoR-15F questionnaire postoperatively
* Subject who has not expressed his opposition to the reuse of his data for scientific research purposes.

Exclusion criteria:

- Subject who expressed their opposition to participating in the study has

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient aged ≥18 years underwent osteoarticular surgery between 01/01/2019 and 31/12/2022.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-01-08 (Estimated); Study Completion 2024-01-08 (Estimated)

PRIMARY OUTCOMES:
Score measurement of the QoR-15F questionnaire | Score measured on D1, D3, D14 and D28 postoperatively
  This conditional probability will be based on the score measurement of the QoR-15F questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eric NOLL, MD, PhD, Principal Investigator — Service d'Anesthésiologie - Réanimation Chirurgicale - CHU de Strasbourg - France
Locations (1):
- Service d'Anesthésiologie - Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France